CLINICAL TRIAL: NCT00862615
Title: Chronic Micro-inflammation and Bone and Muscular Status in Elderly
Brief Title: Relationships Between Quality of Ageing and Age-related Degenerated Disease (Compalimage)
Acronym: Compalimage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Noël CANO, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-0048; IDRCB 2008-A00593-52; AU750
Record Dates: First submitted 2009-03-12; First posted 2009-03-17 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Age-related Degenerated Disease
Keywords: Ageing; Inflammation; Muscle protein synthesis; Osteopenia; Sarcopenia
MeSH Terms: conditions — Inflammation; Bone Diseases, Metabolic; Sarcopenia

INTERVENTIONS:
Other: Measurement of muscle protein synthesis using stable isotopes and muscle biopsies. — Measurement of muscle protein synthesis using stable isotopes and muscle biopsies.
  Isotopes are :
  (13C)bicarbonate (0.09 mg/kg fat-free mass) and L(1-13C)leucine (1.3 mg/kg fat-free mass) (intravenous way) L-(5,5,5 2H3) leucine(0.09 µmoles/(kg de fat-free mass.min) (oral way)

SUMMARY:
This project aims to assess the impact of chronic micro-inflammation on age-related loss of muscle (sarcopenia) and bone (osteopenia). The hypothesis is that chronic micro-inflammation and oxidative stress, which prevalence increases during ageing, may participate in the pathogenesis of both sarcopenia and osteopenia.

DETAILED DESCRIPTION:
In order to explore the effect of a moderate chronic inflammation on skeletal muscle function and protein metabolism and on bone status, two groups of 16 subjects each will be selected according to their inflammatory status ie non-inflamed versus micro-inflamed. The volunteers will be sampled twice at week 0 and week 6 in order to quantify plasma concentration of C reactive protein (CRP) using the ultra sensitive assay. The subjects exhibiting CRP lower than 1 mg/l twice will be included in the non-inflamed group and the subjects exhibiting CRP higher than 3 and lower than 15 mg/l will be included in the micro-inflamed group.

During the two weeks before the metabolic studies dietary intakes, DEXA, muscle function, VO2 max and biomarkers of bone remodelling will be assessed. Volunteers will then be submitted to a diet controlled for its protein content, for 4 days (1 g protein/kg/day and 30 kcal/kg/day) before metabolic investigations. One day before, urine will be collected for metabolomics. On the day of metabolic investigations, after an overnight fast, blood samples will be collected for albumin, fibrinogen, inflammatory cytokine and adipokine determination. Then, the subjects will be perfused with L-[1-13C] leucine for 8 hours (post absorptive sate then post prandial satte) during which expired gas and blood samples will be taken, as well as 2 muscle biopsies. Isotopic enrichments in expired gas, in plasma cetoiscaproate and in free or protein-bound leucine in muscle will be measured to determine proteolysis and proteosynthesis rate of muscle proteins.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Body mass index 21 BMI 30 kg/m2
* Affiliated to National Health Insurance
* Subject giving his written informed consent
* Subject considered as normal after clinical examination and medical questionnaire.

Exclusion Criteria:

* Positive serologies to HIV or HCV, determined on blood samples
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Chronic pathologies : Diabetes, cardiovascular diseases, cancer, chronic inflammation diseases, renal, pulmonary impairments Reported xylocaïne allergy
* Osteoporosis
* Prostate hypertrophy
* Glaucoma
* Heavy consumer of alcohol
* Practising intensive physical exercise
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Dietary habits unreliable to controlled food intake
* Being in exclusion on the National Volunteers Data file

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Isotopic enrichments in expired gas, in plasma cetoisocaproate and in free or protein-bound leucine in muscle will be measured to determine proteolysis and proteosynthesis rate of muscle proteins. | at week 0 and week 6

SECONDARY OUTCOMES:
Splanchnic extraction of amino acids, bone metabolism, muscular strength, global metabolism and quality of life. | at week 0 and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Noël CANO, Principal Investigator — University Hospital, Clermont-Ferrand; Dominique Dardevet, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France